CLINICAL TRIAL: NCT03726892
Title: Comparison of MECHANISM of Early and Late Vascular Responses Following Treatment of ST-elevation Acute Myocardial Infarction With Two Different Everolimus-eluting Stents: Randomized Controlled Trial Between Biodegradable Polymer and Durable Polymer Stent
Brief Title: Comparison of MECHANISM of Early and Late Vascular Responses Following Treatment of ST-elevation Acute Myocardial Infarction With Two Different Everolimus-eluting Stents: Randomized Controlled Trial Between Biodegradable Polymer and Durable Polymer Stent (MECHANISM-AMI-RCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Iwate Medical University (Other)
Responsible Party: Principal Investigator, Yoshihiro Morino, Professor, Iwate Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IwateMedicalU
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The SYNERGY stent (Active Comparator)
  Interventions: Device: PCI
- Xience (Active Comparator)
  Interventions: Device: PCI

INTERVENTIONS:
Device: PCI — Coronary Intervention

SUMMARY:
To place two different everolimus-eluting stents (EES), a bioabsorbable polymer EES (Synergy®) and a permanent-type polymer EES (Xience®), randomly to the ST-elevation acute myocardial infarction (AMI) and to observe and compare the early and chronic vascular responses using the frequency domain optical coherence tomography (FD-OCT). The primary endpoint is the 2-week strut coverage rate by FD-OCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with new coronary lesion indicated for PCI using DES
2. Patients whose age at acquisition of consent is 20 to less than 85 years
3. Patients who themselves or whose representatives showed the written consent
4. Patients who will undergo cardiac catheterization 2 weeks later (staged PCI on the other vessel or confirmatory angiography at the treated site)

Exclusion Criteria:

If the following exclusion criteria are satisfied, the patient should not be enrolled in this study even after acquisition of patient's consent:

1. When the follow-up after 12 months is considered difficult (the patient's residence should also be considered)
2. When there is no obvious ACS finding in angiography (decisions should be left to operator)
3. Patients with shock
4. Patients whose culprit lesion is the left main coronary trunk
5. Lesion with the reference vascular diameter of <2.0 mm or ≥4.5 mm visually
6. AMI that occurred newly at the site where a stent has already been placed
7. Chronic renal failure in which the serum creatinine concentration at visit is ≥2.0 mg/dL
8. Patients undergoing hemodialysis
9. Tumor-bearing patients whose life prognosis is expected to be within 2 years
10. Patients for whom the surgical operation requiring withdrawal of antiplatelet drug is scheduled within 3 months
11. Female patients during pregnancy or scheduled to be pregnant
12. Patients with a past history of the side effect of aspirin, clopidogrel or prasugrel (when the patient is confirmed for the safety of ticlopidine, this does not apply even if there is the side effect of clopidogrel or prasugrel)

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
2-weeks strut coverage rate by FD-OCT | 2-weeks
  In this clinical study, the 2-week covered strut rate by FD-OCT should be considered the primary endpoint, and the non-inferiority of Synergy® to the present standard treatment, Xience®, established in the control group in the treatment of STEMI, should be demonstrated.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiro Morino, MD, Principal Investigator — Iwate Medical University
Locations (1):
- Iwate Medical University Hospital, Morioka, Japan